CLINICAL TRIAL: NCT06781879
Title: Chemoablation Or Bladder Resection With Adjuvant Chemotherapy in Recurrent Non-Muscle Invasive Bladder Cancer
Acronym: COBRA-NMIBC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jakob Kristian Jakobsen (Other)
Collaborators: medac GmbH (Industry); Danish Cancer Society (Other)
Responsible Party: Sponsor-Investigator, Jakob Kristian Jakobsen, Senior consultant and acting head of urological research unit, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COBRA NMIBC
Record Dates: First submitted 2025-01-14; First posted 2025-01-17 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Non-Muscle Invasive Bladder Cancer
Keywords: Recurrence; Ta low.grade; Chemoablation
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Recurrence | interventions — Mitomycin

STUDY DESIGN:
Intervention Model Description: international multicenter RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chemoablation (Experimental): Patients will undergo dose dense chemoablation with MMC three times per week for two weeks (six instillations in total) followed by flexible cystoscopy eight weeks later. If no tumour can be identified (complete response), patients will receive monthly MMC maintenance instillations for 6 months (six instillations in total) and then continue in the outpatient follow-up programme, according to European guidelines. If tumour regression is observed without complete response or there is no response, a TURBT or outpatient biopsy and tumour fulguration will be performed followed by adjuvant BCG with induction therapy and 1 year maintenance (6 weekly instillations as induction followed by 3 weekly instillations as maintenance at 3, 6, and 12 months or 4, 8 and 12 months as is standard for site ).
  Interventions: Drug: Mitomycin c
- Control (No Intervention): Patients will have TURBT or outpatient biopsy and tumour fulguration performed, followed by standard intravesical instillation therapy according to tumour histology: MMC once a week for six weeks with a monthly maintenance instillation for six months in low-grade tumours. For high-grade tumours BCG will be utilised once a week for six weeks followed by 1-year maintenance consisting of one weekly instillation for three weeks after 3, 6, and 12 months or 4, 8 and 12 months as is standard for site.

INTERVENTIONS:
Drug: Mitomycin c — Chemoablation
  Arms: Chemoablation

SUMMARY:
The investigartors will conduct a randomized, multinational study with the aim to assess if the efficacy of a dose dense chemoablation with Mitomycin C (MMC) with adjuvant BCG in non-responding patients is superior regarding long term effect compared to standard treatment with trans urethral resection of bladder tumors (TURBT) and adjuvant intravesical instillation therapy in patients with recurrent Ta LG tumors.

The study is a natural follow-up study following the pivotal NICSA trial supported by the Danish Cancer Society that has lead to the initial change in the European guidelines. In order to not only be comparable to current standard, but also to improve clinical outcome and furthermore confirm the previous findings, the investigators here suggest to implement at patient tailored approach through a new multicenter RCT.

The investigators hypothesize that chemoablation with MMC in patients with recurrent Ta LG tumors will result in a permanent low recurrence rate in patients with complete response, whereas patients without complete response can be selected for adjuvant BCG which theoretically is more efficient in this select patient group. This will potentially result in a more favorable long term recurrence free survival (RFS) rate compared to the current standard regimen where all patients are treated with TURBT and adjuvant instillation therapy.

The incidence of bladder cancer in Denmark is almost 2,000 per year. Of these, 75% have non-muscle invasive bladder cancer (NMIBC). The yearly recurrence rate of NMIBC is approximately 35% and the disease is therefore one of the most costly cancers to manage on a per patient basis, due to the cost of operative procedures, follow-up cystoscopies and instillation therapies

ELIGIBILITY:
Inclusion Criteria:

* Tumour recurrence after previous urothelial tumour of Ta low-grade
* Tumours smaller than 2 cm in diameter
* Negative urine cytology (optional)
* ≥18 years of age
* Ability to understand and comprehend the provided written and oral information
* Has provided written consent

Exclusion Criteria:

* Known history of invasive tumour of the bladder (T1+)
* Known history of CIS of the bladder
* Previous MMC or BCG-treatment except for single instillations following previous TURBTs
* Known allergy or intolerance to MMC
* Solid tumour with suspicions of invasion
* Tumour in the bladder neck or urethra
* Suspicion of CIS (positive cytology with high-grade neoplastic cells combined with suspicious flat lesions seen at cystoscopy)
* Small bladder volume (less than 100 ml) or incontinence
* Prior radiation therapy to the pelvic area, as radiation affects the bladder function and instillation therapy is a suboptimal treatment for this patient group
* Acute cystitis
* Pregnancy or breast-feeding
* Averse to using secure contraception with regard to men with partners and premenopausal women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
Two-year Recurrence Free Survival | 2 years
  This is defined as event of first recurrence following treatment but not including the recurrence diagnosed at the time of inclusion or persisting tumour following chemoablation.

SECONDARY OUTCOMES:
Five-year RFS | 5 years
  This is defined as event of first recurrence following treatment but not including the recurrence diagnosed at the time of inclusion or persisting tumour following chemoablation.
Number of patients in need of a TURBT or tumour fulguration in the outpatient clinic in the first two years following randomisation | 2 years
  need for TURBT/fulgaration
Number of tumours at first recurrence based on the following intervals: 1, 2-7, > 8 | 5 years
  tumour number
Number of TURBTs per patient in the first two and five years of follow-up based on the following intervals: 1, 2-5, 5-10 and multiple | 5 years
  number of TURBTs
Five-year progression free survival | 5 years
  (progression defined as progression to T1-tumour, T2+-tumour, or cystectomy irrespectively of indication)
Five-year overall survival | 5 years
  survival
Number of patients completing assigned intervention | 2 years
  completing assigned intervention
Serious adverse events related to MMC treatment during neoadjuvant or adjuvant therapy | 2 years
  SAE's

CONTACTS AND LOCATIONS:
Locations (8):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Herlev and Gentofte Hospital, Herlev
  - Zealand University Hospital, Roskilde, Roskilde
- Landspítali University Hospital, Reykjavik, Iceland
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Vestfold Hospital Trust, Tønsberg
- NU Hospital Group, Uddevalla, Sweden

IPD SHARING:
Plan to Share IPD: No